CLINICAL TRIAL: NCT04947566
Title: Comparison of Efficacy of Naproxen Versus Ibuprofen in the Management of Post-Operative Endodontic Pain in Teeth With Irreversible Pulpitis
Brief Title: Comparison of Efficacy of Naproxen Versus Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, Zarlashta Usman, ZUsman, Fatima Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZUsman
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naproxen (Experimental): in this group patients were given Naproxen
  Interventions: Drug: Comparison of Efficacy of Naproxen versus Ibuprofen
- Ibuprofen (Experimental): in this group patients were given ibuprofen
  Interventions: Drug: Comparison of Efficacy of Naproxen versus Ibuprofen

INTERVENTIONS:
Drug: Comparison of Efficacy of Naproxen versus Ibuprofen — Comparison of Efficacy of Naproxen Versus Ibuprofen in the Management of Post-Operative Endodontic Pain in Teeth with Irreversible Pulpitis

SUMMARY:
Comparison between Naproxen and Ibuprofen in management of post operative endodontic pain was done.Total 116 patients were selected and divided in to two groups.One group was given Naproxen and other was given Ibuprofen.

DETAILED DESCRIPTION:
This Randomized Controlled Trial was carried out in Outpatient Department of Operative Dentistry, Fatima Memorial Hospital, Lahore, Pakistan and was completed in six months from September 2nd,2019 to February 25th,2020. Sample size of 116 cases(58 in each group) of irreversible pulpitis was calculated with 80% power of test, 5% level of significance, P1(prevalence) for naproxen was 61.53% and P2 for ibuprofen is 38.46%. Estimation of P (prevalence) as 90% is based on pilot study carried in our Department. The patients were randomly allocated into two groups, A and B, by random number table. In both groups teeth were anaesthetized using 1.8ml of 2% lignocaine containing 1:100,000 epinephrine and isolated with rubber dam. An access cavity was prepared with round bur and pulpectomy was done using hand files. Working length was determined using an electronic apex locator and confirmed with periapical radiograph. Canals were prepared with step back technique. Canals were then dried with paper points and the access cavities were restored temporarily with cavit(Cavit3M ESPE).Visual analogue scale for pain score was measured for both groups before initial endodontic procedure . group A was given (naproxen 550 mg B.D), while group B was given (Ibuprofen 400mg B.D).Post-operative pain was measured subjectively after 24 hours with standard Visual Analogue Score (VAS) scored on a 10 cm scale, with markings at every 1 cm anchored by the end points of "no pain" on the left and "worst pain" on the right. Patient were asked to point the number most precisely describing the amount of pain he or she experienced after 24 hours. All this data was recorded in a specially designed proforma (attached).Efficacy was labelled as per operational definitions. Data was analyzed using SPSS version 20. For descriptive analysis, mean and standard deviation were reported for age, BMI and VAS score, whereas frequency and percentages were calculated for categorical variables like gender and educational status. A chi square was used to determine the significance of the difference between the efficacy of naproxen and ibuprofen. Data was stratified for age, gender, BMI and educational status .This comparison also included feelings of patients in terms of side effects. A p value 0.05 or less was taken as significant. Post stratification chi-square was applied with p value ≤0.05 considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* • Age range 20-40 years

  * Gender- either
  * Teeth with acute Irreversible pulpitis assessed by Electric pulp tester lasting more than 30 seconds
  * One tooth per arch with no opposing tooth involved

Exclusion Criteria:

* Patients who reported to have any systemic disease while taking history e.g. diabetes, hypertension
* During pregnancy
* History of taking analgesics 12 hours prior to treatment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
post-operative pain | 6 months
  Post-operative pain was measured subjectively after 24 hours with standard Visual Analogue Score (VAS) scored on a 10 cm scale, with markings at every 1 cm anchored by the end points of "no pain" on the left and "worst pain" on the right. Patient were asked to point the number most precisely describing the amount of pain he or she experienced after 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Zarlashta Usman, BDS, Principal Investigator — Fatima Memorial Hospital
Locations (2):
- Pakistan (2):
  - FatimaMH, Lahore, Punjab Province
  - FatinaMH, Lahore, Punjab Province